CLINICAL TRIAL: NCT01942317
Title: The Role of Balneotherapy in Obese Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Stefano Masiero, Professore Ordinario, University of Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20232; 20232; 20232 (Other: COMITATO ETICO PER LA SPERIMENTAZIONE - AZIENDA OSPEDALIERA DI PADOVA, ITALY)
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Knee Osteoarthritis, Obesity
MeSH Terms: conditions — Osteoarthritis, Knee; Obesity | interventions — Balneology

ARMS (2):
- Balneotherapy (Experimental): 16 balneotherapy treatments, each of 45 minutes, twice a week, for 8 consecutive weeks
  Interventions: Other: Balneotherapy
- Physiotherapy (No Intervention): 16 physiotherapy treatments (no balneotherapy), each of 45 minutes, twice a week, for 8 consecutive weeks

INTERVENTIONS:
Other: Balneotherapy
  Arms: Balneotherapy

SUMMARY:
The aim of the study is to evaluate the role of balneotherapy in obese patients with knee osteoarthritis in terms of pain relief, improving joint function and deambulation, on endocrinological parameters, quality of life and of reduction the costs to "Servizio Sanitario Nazionale" (NHS).

ELIGIBILITY:
Inclusion Criteria:

* obesity II-III grade (BMI 35-45 kg/m2)
* knee pain
* patient compliance to the treatment

Exclusion Criteria:

* BMI<34,9kg/m2 or BMI> 45,1kg/m2
* previous knee surgery
* complicated diabetes mellitus
* ischemic cardiomyopathy and heart failure
* acute phase of osteoarthritis
* varicose veins, deep venous thrombosis (DVT)
* cancer
* cutaneous lesions
* NSAIDs administration <1 week before the treatment
* knee infiltration <2 months before the treatment

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-03 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Knee pain measurement with Visual Analogue Scale (VAS) | At the begining and at the end of the treatment. After 6 months of the end of therapy

SECONDARY OUTCOMES:
Knee range of motion | At the begining and at the end of the treatment. After 6 months of the end of therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera-Università degli studi di Padova, Padua, Italy, Italy